CLINICAL TRIAL: NCT01932398
Title: Posterior Alpha Oscillations as an Index for the Attentional Bias in Children With Attentional Deficit Hyperactivity Disorder
Brief Title: A Study on the Inter-Hemispheric Alpha Ratio in Kids With ADHD (SHARK)
Acronym: SHARK
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 3016038.01
Record Dates: First submitted 2013-08-22; First posted 2013-08-30 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: ADHD
Keywords: Alpha; Lateralization; Attention; ADHD; Oscillation
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ADHD: A diagnosis of ADHD, classified by the DSM-IV.
- no ADHD: No diagnosis of ADHD, classified by the DSM-IV.

SUMMARY:
Investigate the hypothesis that children with ADHD have difficulty with the allocation of visio-spatial attention related to an inability to control posterior alpha brain oscillations. A paradigm will be used in which the aim is to address covert attention as similar recent studies did in adults with ADHD.

ELIGIBILITY:
Inclusion Criteria:

For both groups

* Age between 7 and 10 years of age.
* Estimated IQ above 80.
* Psychopharmaca- naïve or -free.

For the ADHD-group - A diagnosis of ADHD, classified by the DSM-IV.

Exclusion Criteria:

* (Co-morbid) psychiatric disorder (major depression, bipolar disorder, psychotic disorder, chronically motor tic disorder or Gilles de la Tourette, Conduct disorder, autism spectrum disorder, eating disorder, anxiety disorder).
* Neurological disorders (e.g. epilepsy) currently or in the past.
* Cardiovascular disease currently or in the past.
* Serious motor or perceptual handicap.

For the no ADHD-group

- No diagnosis of ADHD, classified by the DSM-IV.

Ages: 84 Months to 95 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: ADHD vs no ADHD
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Modualtion of alpha power | Once for half an hour
  Modulation* of alpha power on congruent and incongruent trials of the covert attention task in 30 ADHD children and in 30 non-ADHD children
  *Modulation is the (expected) cue-induced change by a covert attention task.

SECONDARY OUTCOMES:
Response time on covert attention task | Once for half an hour
  Time it takes to press the correct button after presentation of target-stimulus on congruent and incongruent trials of the covert attention task in 30 ADHD children and 30 non-ADHD children
Standard deviation of response time on covert attention task | Once for half an hour
  The variation of the time it takes to press the correct button after presentation of target-stimulus on congruent and incongruent trials of the covert attention task in 30 ADHD children and 30 non-ADHD children
Correct responses on covert attention task | Once for half an hour
  Number of correct button presses responses (i.e. same side as the target) on the covert attention task on congruent and incongruent trials of the covert attention task in 30 ADHD children and 30 non-ADHD children
Mean deviation from middle on line bisection task | Once in about 5 minutes
  Mean deviation in mm from the center of the line on the line bisection task for 30 ADHD children and 30 non-ADHD children
Inattention score on the ADHD-RS-IV | Once in about 10 minutes
  The inattention subscale of the ADHD-RS-IV for 30 ADHD children and 30 non-ADHD children
Hyperactivity/impulsivity score on the ADHD-RS-IV | Once in about 10 minutes
  The hyperactivity/impulsivity subscale of the ADHD-RS-IV for 30 ADHD children and 30 non-ADHD children

OTHER OUTCOMES:
FSIQ estimation | Once in about 20 minutes
  An estimate of full scale IQ, measured with 2 subtests of the WISC-III for 30 ADHD-children and 30 non-ADHD children

CONTACTS AND LOCATIONS:
Overall Officials: Ole Jensen, Prof, Principal Investigator — Donders Institute for Brain, Cognition and Behavior - Centre for Cognitive Neuroimaging; Jan K Buitelaar, Prof, Principal Investigator — Radboud University, Medical Centre - Donders Institute for Brain, Cognition and Behavior, Department of Cognitive Neuroscience
Locations (1):
- Donders Institute for Brain, Cognition and Behavior, Centre for Cognitive Neuroimaging, Nijmegen, Gelderland, Netherlands